CLINICAL TRIAL: NCT02063360
Title: Open-Label, Single-Sequence Study to Evaluate the Pharmacokinetic Interaction of BMS-663068 With Darunavir/Ritonavir and/or Etravirine in Healthy Subjects
Brief Title: DDI Study of BMS-663068 With Etravirine (ETR) and/or Darunavir (DVR) + Ritonavir (RTV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 206281; AI438-020 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir; Darunavir; Ritonavir; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: BMS-663068+DRV/RTV (Experimental): Extended release tablet BMS-663068 600mg orally twice daily on days 1-4 and 17-26. Tablet DRV 600mg / RTV 100mg orally orally twice daily on days 7-16
  Interventions: Drug: BMS-663068; Drug: Darunavir (DRV); Drug: Ritonavir (RTV)
- Cohort 2: BMS-663068+ETR (Experimental): Extended release tablet BMS-663068 600mg orally twice daily on days 1-4 and 17-26. Tablet ETR 200mg orally orally twice daily on days 7-16
  Interventions: Drug: BMS-663068; Drug: Etravirine (ETR)
- Cohort 3: BMS-663068+DRV/RTV+ETR (Experimental): Extended release tablet BMS-663068 600mg orally twice daily on days 1-4 and 17-26. Tablet DRV 600mg / RTV 100mg and ETR 200mg orally orally twice daily on days 7-16
  Interventions: Drug: BMS-663068; Drug: Darunavir (DRV); Drug: Ritonavir (RTV); Drug: Etravirine (ETR)

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068
Drug: Darunavir (DRV) — Darunavir (DRV)
  Other Names: Prezista
  Arms: Cohort 1: BMS-663068+DRV/RTV; Cohort 3: BMS-663068+DRV/RTV+ETR
Drug: Ritonavir (RTV) — Ritonavir (RTV)
  Other Names: Norvir
  Arms: Cohort 1: BMS-663068+DRV/RTV; Cohort 3: BMS-663068+DRV/RTV+ETR
Drug: Etravirine (ETR) — Etravirine (ETR)
  Other Names: Intelence
  Arms: Cohort 2: BMS-663068+ETR; Cohort 3: BMS-663068+DRV/RTV+ETR

SUMMARY:
The purpose of this study is to determine if there is an interaction in healthy subjects taking BMS-663068 with Darunavir/Ritonavir and/or Etravirine.

DETAILED DESCRIPTION:
Brief title: drug-drug interaction (DDI)

Primary Purpose: Other : Phase 1 Clinical Pharmacology drug interaction study in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no clinically significant deviation from normal in medical history, physical examination findings, 12-lead ECG measurements, and clinical laboratory tests
* Women of childbearing potential (WOCBP) allowed. Must be practicing highly effective methods of contraception

Exclusion Criteria:

* Any significant acute or chronic medical condition
* Unable to tolerate oral medications
* Inability to be venipunctured and/or tolerate venous access
* Current or recent (within 3 months of dosing) gastrointestinal disease
* Abnormal liver function test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02-01; Primary Completion 2014-05-01 (Actual); Study Completion 2014-05-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-626529 | 20 timepoints up to day 26
Area under the concentration-time curve in 1 dosing interval (AUC(TAU)) of BMS-626529 | 20 timepoints up to day 26

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) for BMS-626529, DRV, RTV, and ETR | Up to day 26 (20 timepoints for BMS-626529, 24 timepoints for DRV, RTV and ETR)
Concentration at 12 hours (C12) for BMS-626529, DRV, RTV, and ETR | Up to day 26 (20 timepoints for BMS-626529, 24 timepoints for DRV, RTV and ETR)
Trough observed plasma concentration (Ctrough) for BMS-626529, DRV, RTV, and ETR | Up to day 26 (20 timepoints for BMS-626529, 24 timepoints for DRV, RTV and ETR)
Cmax for DRV, RTV, and ETR | 24 timepoints up to 26 day
AUC(TAU) for DRV, RTV, and ETR | 24 timepoints up to 26 day
Safety and tolerability endpoints include incidence of adverse event (AEs), serious adverse event (SAEs), AEs leading to discontinuation, deaths, marked laboratory abnormalities, and abnormalities in vital signs, physical examination, and 12-lead ECGs | Up to day 27

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare

REFERENCES:
- [Derived] Moore K, Thakkar N, Magee M, Sevinsky H, Vakkalagadda B, Lubin S, Llamoso C, Ackerman P. Pharmacokinetics of Temsavir, the Active Moiety of the HIV-1 Attachment Inhibitor Prodrug, Fostemsavir, Coadministered with Cobicistat, Etravirine, Darunavir/Cobicistat, or Darunavir/Ritonavir with or without Etravirine in Healthy Participants. Antimicrob Agents Chemother. 2022 Apr 19;66(4):e0225121. doi: 10.1128/aac.02251-21. Epub 2022 Mar 22. PMID 35315687